CLINICAL TRIAL: NCT04761211
Title: Effect and Safety of Smart Bra of Peking Union Medical College & Hospital
Brief Title: Effect and Safety of Smart Bra (PUMCH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCH-ESSB
Record Dates: First submitted 2020-09-02; First posted 2021-02-18 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Effects of the Elements
Keywords: effectiveness; safety; smart bra

STUDY DESIGN:
Intervention Model Description: The patients who were going to receive double breast ultrasound and molybdenum target in the breast surgery clinic and ward were enrolled into the group (disease-free: benign: malignant = 1:1:1). The patients were put on the device for about 3 minutes, and the breast was photographed at 5 sites. After that, the artificial intelligence learning was carried out on the photos of the training group. For the photos of the verification group, the algorithm obtained by the training group was compared with the existing artificial intelligence algorithms of ultrasound and molybdenum target.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- smart bra (Experimental): The patients who were going to take breast ultrasound in the breast surgery clinic were enrolled into the group. The patients were put on the device for about 3 minutes, and the breast was photographed at 5 sites. After that, the artificial intelligence learning was carried out on the photos of the training stage. For the photos of the verification stage, the algorithm obtained by the training stage was compared with the existing artificial intelligence algorithms of ultrasound and molybdenum target.
  Interventions: Device: smart bra

INTERVENTIONS:
Device: smart bra — This is a patented infrared breast examination bra

SUMMARY:
This is a multicenter, prospective clinical study was conducted to evaluate the safety and effectiveness of Xiehe smart bra for breast disease screening in outpatients with breast surgery. According to the patients' wishes and written informed consent, they were randomly assigned to the study group. A total of 2000 patients were expected to be enrolled. The training group: validation group = 1:1.

DETAILED DESCRIPTION:
This study is a randomized, open, multicenter clinical study. It will be conducted in Peking Union Medical College Hospital, Shanxi Provincial People's Hospital, Beijing Third Hospital, Zhalantun ZhongMeng hospital, Chongqing Medical University affiliated university town hospital, Shenzhen People's Hospital and other national hospitals. A total of 2000 subjects are expected to participate. The patients in the group wore the device for about 3 minutes, and took photos of 5 breast sites. After that, the artificial intelligence learning was carried out on the photos of the training group. For the photos of the verification group, the algorithm obtained by the training group was compared with the existing artificial intelligence algorithms of ultrasound and molybdenum target. During the follow-up, the safety of the product was evaluated. According to the basic principles of safety and performance of who international general GHTF (sg1-n020r5) medical devices.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are going to receive breast ultrasound and molybdenum target in breast surgery clinic;
2. Female patients (18-80 years old);
3. Signed written informed consent approved by the relevant institutional review board (IRB) or independent ethics committee (IEC)

Exclusion Criteria:

1. The subjects were pregnant or lactating;
2. Patients with nipple discharge;
3. Known allergy to bra materials;
4. The patients who had received breast surgery or breast puncture within half a year;
5. Patients with skin diseases.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2141 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity | baseline
  Using ultrasound and / or pathological results as the gold standard, the positive rates of breast diseases (benign breast diseases and malignant breast diseases) detected by smart bra are recorded.

SECONDARY OUTCOMES:
Specificity | baseline
  Using ultrasound and / or pathological results as the gold standard, the probability of no breast disease (benign breast disease, malignant breast disease) are recorded

OTHER OUTCOMES:
Number of adverse events assessed by CTCAE v4.0 | baseline; 3months
  Number of participants with smart-bra related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Xuefei Wang, Study Chair — PUMCH
Locations (1):
- Breast Surgery Department of PUMCH, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
We will decide during this trial.

REFERENCES:
- [Derived] Wang X, Chou K, Zhang G, Zuo Z, Zhang T, Zhou Y, Mao F, Lin Y, Shen S, Zhang X, Wang X, Zhong Y, Qin X, Guo H, Wang X, Xiao Y, Yi Q, Yan C, Liu J, Li D, Liu W, Liu M, Ma X, Tao J, Sun Q, Zhai J, Huang L. Breast cancer pre-clinical screening using infrared thermography and artificial intelligence: a prospective, multicentre, diagnostic accuracy cohort study. Int J Surg. 2023 Oct 1;109(10):3021-3031. doi: 10.1097/JS9.0000000000000594. PMID 37678284

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/11/NCT04761211/Prot_SAP_ICF_000.pdf